CLINICAL TRIAL: NCT00545194
Title: Randomized Study on Removable PGE2 Vaginal Insert Versus PGE2 Intravaginal Gel for Cervical Priming and Labour Induction in Term Pregnancy
Brief Title: Cervical Ripening Before Induction of Labour at Term: a Randomised Comparison of Prostin vs Propess
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: PROPESS Study
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2007-10

CONDITIONS: Cervical Ripening; Labor, Induced
Keywords: Prostaglandin E2; Intravaginal gel; Bishop score; Induction of labor; randomized trial; Vaginal insert
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): sustained release preparation of prostaglandin E2
  Interventions: Drug: Prostaglandin E2
- B (Active Comparator): short-acting (instant-released) preparation of prostaglandin E2
  Interventions: Drug: Prostaglandin E2

INTERVENTIONS:
Drug: Prostaglandin E2

SUMMARY:
The aim of this study is to compare two different preparation

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* cephalic presentation
* gestation of more than 37 Weeks confirmed by ultrasound
* Bishop score less than 7
* Informed consent

Exclusion Criteria:

* previous cesarean section (scarred uterus)
* polyhydramnios
* multiple pregnancy
* fetal malformation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2002-01 (Actual); Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Percentage of vaginal deliveries within the 48 hours after cervical ripening | 48 hours

SECONDARY OUTCOMES:
Proportion of total vaginal deliveries | 48 hours
Vaginal deliveries at 12 hours, 24 hours and 36 hours | 48 hours
Number of hyperkinesia with or without fetal heart rate monitoring abnormalities | 48 hours
Number of hypertonia with or without fetal heart rate monitoring abnormalities | 48 hours
Apgar score at 5 min less or equal 7 | 48 hours
Apgar score at 10 min less or equal 7 | 48 hours
Arterial pH less or equal 7.20 | 48 hours
Arterial base excess more than 12 | 48 hours
Number of maternal post-partum haemorrhage | 48 hours
Time to reach 3cm cervical dilatation | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Franck Perrotin, MD-PhD, Principal Investigator — Tours Universiity Hospital
Locations (1):
- Olympe de Gouges Women Health Centre, Bretonneau University Hospital, Tours, France

REFERENCES:
- [Background] Lyrenas S, Clason I, Ulmsten U. In vivo controlled release of PGE2 from a vaginal insert (0.8 mm, 10 mg) during induction of labour. BJOG. 2001 Feb;108(2):169-78. doi: 10.1111/j.1471-0528.2001.00039.x. PMID 11236117
- [Background] Strobelt N, Meregalli V, Ratti M, Mariani S, Zani G, Morana S. Randomized study on removable PGE2 vaginal insert versus PGE2 cervical gel for cervical priming and labor induction in low-Bishop-score pregnancy. Acta Obstet Gynecol Scand. 2006;85(3):302-5. doi: 10.1080/00016340500523685. PMID 16553177
- [Background] El-Shawarby SA, Connell RJ. Induction of labour at term with vaginal prostaglandins preparations: a randomised controlled trial of Prostin vs Propess. J Obstet Gynaecol. 2006 Oct;26(7):627-30. doi: 10.1080/01443610600903362. PMID 17071427